CLINICAL TRIAL: NCT03364751
Title: A 6-month Randomized, Controlled, Open-label, 2-arm Parallel Group, Multicenter Study to Evaluate the Effect of Switching From Cigarette Smoking to the Use of IQOS in Smokers With Generalized Chronic Periodontitis on the Response to Mechanical Periodontal Treatment and Oral Health Status.
Brief Title: Effect of Switching From Cigarette Smoking to the Use of IQOS on Periodontitis Treatment Outcome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philip Morris Products S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: P1-OHS-01-JP
Record Dates: First submitted 2017-11-23; First posted 2017-12-07 (Actual); Results first posted 2021-02-18 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Periodontal Diseases; Chronic Periodontitis; Periodontal Pocket; Tooth Mobility; Gingival Diseases; Smoking, Cigarette
Keywords: Oral Health; Smoking; Cigarette; Reduced risk product; Tobacco heating system; THS; Modified risk tobacco product; Clinical attachment level
MeSH Terms: conditions — Periodontal Diseases; Chronic Periodontitis; Periodontal Pocket; Tooth Mobility; Gingival Diseases; Cigarette Smoking; Smoking | interventions — Tobacco Products

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The Dentist (Investigator) or Dental Hygienist performing the periodontal assessments will be blinded to the arm allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IQOS arm (Active Comparator): ~86 patients, switching from cigarette smoking to IQOS use.
  Interventions: Other: IQOS
- Cigarette arm (Active Comparator): ~86 patients, continuing cigarette smoking.
  Interventions: Other: Cigarette

INTERVENTIONS:
Other: IQOS — Patients will switch from cigarette smoking to ad libitum IQOS use.
  Arms: IQOS arm
Other: Cigarette — Patients will continue to smoke cigarettes ad libitum.
  Arms: Cigarette arm

SUMMARY:
The purpose of this study was to demonstrate in patients with generalized chronic periodontitis that switching from cigarette smoking to using IQOS improves the response to periodontal therapy and the overall oral health status compared to continuing cigarette smoking.

Note: "IQOS" is the Tobacco Heating System (THS) with Marlboro Heatsticks, marketed in Japan under the brand name IQOS

DETAILED DESCRIPTION:
This was a randomized, controlled, open-label, 2-arm, parallel group ambulatory study with the randomization stratified by daily cigarette consumption over the month (30 days) prior to Visit 1 (10-19 cigarettes/day vs. > 19 cigarettes/day) and disease severity recorded at Visit 1 (< 5 mm Pocket Depth [PD] vs. ≥ 5 mm PD) based on the most severely diseased tooth, in smokers with generalized chronic periodontitis who are randomized to either switch from cigarette smoking to IQOS use or continuing cigarette smoking.

ELIGIBILITY:
Main Inclusion Criteria:

1. Patient is aged ≥ 30 years old.
2. Patient has smoked on average at least 10 commercially available cigarettes per day for at least 5 years
3. Patient has generalized chronic periodontitis (i.e., more than 30% of diseased teeth with a PD ≥ 4 mm).

Main Exclusion Criteria:

1. Patient has self-reported history of diagnosed systemic diseases (e.g., stroke or acute cardiovascular event within the last 5 years, diabetes, active cancer).
2. Patient received root planing therapy within the 6 months prior to Visit 1.
3. Patient received surgical periodontal therapy within 3 years prior to Visit
4. Patient was treated within the 3 months prior to Visit 1 with systemic antibiotics or was treated with topical antibiotics applied in the mouth.
5. Continuous systemic use of steroidal or non-steroidal anti-inflammatory drugs for more than 20 days during the past 30-day period (except for low dose aspirin, i.e., ≤300 mg).
6. Female patients who are pregnant, breast-feeding, or planning a pregnancy within the course of the study.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2017-11-07 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2019-06-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christelle Haziza, PhD, Study Chair — Philip Morris Products S.A.
Locations (26):
- Japan (26):
  - Mase Dental Clinic, Futtsu, Chiba
  - Tsudanuma Olive Dental Clinic, Narashino, Chiba
  - Matsunobu Dental Office, Miyako, Fukuoka
  - Taniguchi Dental Clinic, Sapporo, Hokkaido
  - Takano Dental Clinic, Chikusei, Ibaraki
  - Tsukuba Healthcare Dental Clinic, Tsukuba, Ibaraki
  - AOI Universal Hospital, Kawasaki, Kanagawa
  - Yoshinaga Dental Office, Uki, Kumamoto
  - Yoshino Dental Clinic, Kawaguchi, Saitama
  - Saida Dental Clinic, Tokorozawa, Saitama
  - Sakai Dental Clinic, Bunkyō, Tokyo
  - Kudan Dental Clinic, Chiyoda City, Tokyo
  - Yano Dental Clinic, Chōfu, Tokyo
  - Nikaido Dental Clinic, Chūō, Tokyo
  - Mune Dental Clinic, Setagaya City, Tokyo
  - Kikuchi Dental Clinic, Shinjuku, Tokyo
  - Miyata Dental Clinic, Toshima City, Tokyo
  - Kato Dental Clinic, Himi, Toyama
  - Kimura Dental Clinic, Fukuoka
  - Yamashita Dental Office, Fukuoka
  - Yasumasu Dental Office, Fukuoka
  - Tsukiyama Dental Clinic, Fukuoka
  - Yoshida Shigeru Dental Office, Fukuoka
  - Yamashita Dental Clinic, Kagoshima
  - Heart Dental Clinic, Kagoshima
  - Higashi Dental Office, Kumamoto

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pouly S, Ng WT, Benzimra M, Soulan A, Blanc N, Zanetti F, Picavet P, Baker G, Haziza C. Effect of Switching to the Tobacco Heating System Versus Continued Cigarette Smoking on Chronic Generalized Periodontitis Treatment Outcome: Protocol for a Randomized Controlled Multicenter Study. JMIR Res Protoc. 2021 Jan 18;10(1):e15350. doi: 10.2196/15350. PMID 33459599
- [Result] Effect of switching from cigarette smoking to the use of the tobacco heating system on periodontitis treatment outcome: Periodontal parameter results from a multicenter Japanese study Authors: Pouly, Sandrine; Ng, Wee Teck; Blanc, Nicolas; Hession, Paul; Zanetti, Filippo; Battey, James N. D.; de La Bourdonnaye, Guillaume; Heremans, Annie; Haziza, Christelle Journal Title: Frontiers in dental medicine Publication Date: 7/22/2022 Volume: 3 DOI: 10.3389/fdmed.2022.915079

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 179 subjects were enrolled in the study. 172 subjects were randomized to the IQOS arm (n=87) or to the cigarette arm (n=85).
  The analysis was performed according to subjects' exposure (Product Use Category, i.e., IQOS; Cigarette; Dual use; or Other) over the study period as detailed in the "Arm/Group" (Reporting Groups) table.
Groups:
- IQOS: IQOS Product Use Category:
  Subjects using over 30 HeatSticks, but less than 30 cigarettes monthly were classified as "IQOS" users (based on self-report).
- Cigarette: Cigarette Product Use Category:
  Monthly users of less than 30 HeatSticks, but over 30 cigarettes were classified as "Cigarette" users (based on self-report).
- Dual User: Dual User Product Use Category:
  Users of over 30 HeatSticks and over 30 cigarettes per month were classified as "Dual User" (based on self-report).
- Other: Other Product Use Category:
  All other use patterns were classified as "Other" (based on self-report).
Period: Overall Study
Arm/Group | IQOS | Cigarette | Dual User | Other
Started | 70 | 84 | 17 | 1
Completed | 69 | 83 | 17 | 1
Not Completed | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Subjects using during the course of this study over 30 HeatSticks, but less than 30 cigarettes monthly were classified as "IQOS" users. Monthly users of less than 30 HeatSticks, but over 30 cigarettes were classified as "Cigarette" users. Users of over 30 HeatSticks and over 30 cigarettes per month were classified as "Dual User". All other use patterns were classified as "Other".
Groups:
- IQOS: IQOS Product Use Category
- Cigarette: Cigarette Product Use Category
- Dual User: Dual User Product Use Category
- Other: Other Product Use Category
- Total: Total of all reporting groups
Arm/Group | IQOS | Cigarette | Dual User | Other | Total
Number analyzed (Participants) | 70 | 84 | 17 | 1 | 172
Age, Continuous [Mean (Full Range); unit: years] | 48.1 [30 to 71] | 46.5 [30 to 77] | 54.4 [33 to 73] | 54.0 [54 to 54] | 48.0 [30 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 17 | 3 | 0 | 33
  Male | 57 | 67 | 14 | 1 | 139
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 70 | 84 | 17 | 1 | 172
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Japan | 70 | 84 | 17 | 1 | 172
Nationality [Count of Participants; unit: Participants]
  Japanese | 70 | 84 | 17 | 1 | 172
  Non-Japanese | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Periodontal Pocket Depth (PD) Change From Baseline at 6 Months
Description: Pocket depth (PD) is the distance from the gingival margin to which a probe penetrates into the pocket. Mean Periodontal PD change from baseline will be measured in all sites with initial PD ≥ 4 mm, following mechanical periodontal therapy, in patients who switch to IQOS use compared to those who continue cigarette smoking.
Time Frame: At 6 months
Population: The analysis population consisted of all randomized subjects with at least one product use experience and at least one valid non-safety assessment. Subjects were analyzed based on their actual self-reported product use. Some participants were excluded from analysis for protocol deviations (including, but not limited to, missing measurements). The "Other" reporting group, which included one subject, was not included in this analysis.
Measure: Mean (95% Confidence Interval); unit: millimeters
Arm/Group | IQOS | Cigarette | Dual User
Number analyzed (Participants) | 70 | 84 | 17
millimeters | -1.046 [-1.194 to -0.898] | -1.114 [-1.258 to -0.970] | -1.177 [-1.399 to -0.956]
Statistical Analysis 1: Comparison: IQOS vs Cigarette; Month 6: Difference between Cigarette and IQOS; Test type: Other; p = 0.297, Mixed Models Analysis; LS Mean Difference = 0.068, 95% CI 2-sided [-0.060 to 0.196]
Statistical Analysis 2: Comparison: Cigarette vs Dual User; Month 6: Difference between Cigarette and Dual Use; Test type: Other; p = 0.550, Mixed Models Analysis; LS Mean Difference = -0.064, 95% CI 2-sided [-0.273 to 0.146]

2. Secondary Outcome: Periodontal Pocket Depth (PD) Change Over Time. (Mean PD in All Subjects With Initial PD ≥ 4 mm)
Description: as for outcome 1
Time Frame: At 3 months
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: millimeters
Groups:
- IQOS: IQOS Product Use Category - As Exposed Set
- Cigarette: Cigarette Product Use Category - As Exposed Set
- Dual User: Dual User Product Use Category - As Exposed Set
Arm/Group | IQOS | Cigarette | Dual User
Number analyzed (Participants) | 70 | 84 | 17
millimeters | -0.972 [-1.120 to -0.824] | -1.016 [-1.158 to -0.873] | -1.035 [-1.257 to -0.814]
Statistical Analysis 1: Comparison: IQOS vs Cigarette; Month 3: Difference between Cigarette and IQOS; Test type: Other; p = 0.502, Mixed Models Analysis; LS Mean Difference = 0.043, 95% CI 2-sided [-0.084 to 0.171]
Statistical Analysis 2: Comparison: Cigarette vs Dual User; Month 3: Difference between Cigarette and Dual Use; Test type: Other; p = 0.851, Mixed Models Analysis; LS Mean Difference = -0.020, 95% CI 2-sided [-0.229 to 0.189]

3. Secondary Outcome: Clinical Attachment Level (CAL) Change Over Time (Mean CAL in All Subjects With Initial PD ≥ 4 mm)
Description: Clinical attachment level (CAL) is the measured distance from cementoenamel junction (CEJ) to the bottom of pocket using a periodontal probe. Mean CAL change from baseline will be measured in sites with initial PD ≥ 4 mm, following mechanical periodontal therapy, in patients who switch to IQOS use compared to those who continue cigarette smoking.
Time Frame: At 3 months and 6 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: millimeters
Arm/Group | IQOS | Cigarette | Dual User
Number analyzed (Participants) | 70 | 83 | 17
millimeters
  Month 3: Change from Baseline | -0.820 [-0.980 to -0.660] | -0.889 [-1.043 to -0.736] | -0.865 [-1.122 to -0.608]
  Month 6: Change from Baseline: number analyzed (Participants) | 69 | 82 | 17
  Month 6: Change from Baseline | -0.903 [-1.064 to -0.743] | -0.995 [-1.150 to -0.840] | -1.100 [-1.357 to -0.843]
Statistical Analysis 1: Comparison: IQOS vs Cigarette; Month 3: Difference between Cigarette and IQOS; Test type: Other; p = 0.376, Mixed Models Analysis; LS Mean Difference = 0.070, 95% CI 2-sided [-0.085 to 0.224]
Statistical Analysis 2: Comparison: Cigarette vs Dual User; Month 3: Difference between Cigarette and DualUse; Test type: Other; p = 0.848, Mixed Models Analysis; LS Mean Difference = 0.025, 95% CI 2-sided [-0.229 to 0.279]
Statistical Analysis 3: Comparison: IQOS vs Cigarette; Month 6: Difference between Cigarette and IQOS; Test type: Other; p = 0.246, Mixed Models Analysis; LS Mean Difference = 0.092, 95% CI 2-sided [-0.064 to 0.247]
Statistical Analysis 4: Comparison: Cigarette vs Dual User; Month 6: Difference between Cigarette and Dual Use; Test type: Other; p = 0.417, Mixed Models Analysis; LS Mean Difference = -0.105, 95% CI 2-sided [-0.359 to 0.150]

4. Secondary Outcome: Periodontal Pocket Depth (PD) Change Over Time. (Mean PD in All Subjects With Initial PD ≥ 4 mm) - Descriptive Statistics
Description: as for outcome 1
Time Frame: From baseline to 3 months and 6 months
Population: The analysis population consisted of all randomized subjects with at least one product use experience and at least one valid non-safety assessment. Subjects were analyzed based on their actual self-reported product use. Some participants were excluded from analysis for protocol deviations (including, but not limited to, missing measurements).
Measure: Least Squares Mean (95% Confidence Interval); unit: millimeters
Arm/Group | IQOS | Cigarette | Dual User | Other
Number analyzed (Participants) | 70 | 84 | 17 | 1
millimeters
  Baseline | 4.45 [4.34 to 4.56] | 4.43 [4.35 to 4.51] | 4.34 [4.25 to 4.44] | 4.07
  Month 3 | 3.44 [3.28 to 3.60] | 3.47 [3.34 to 3.60] | 4.34 [4.25 to 4.44] | 3.04
  Month 6: number analyzed (Participants) | 69 | 83 | 17 | 1
  Month 6 | 3.36 [3.20 to 3.52] | 3.37 [3.23 to 3.51] | 3.29 [3.03 to 3.54] | 3.09

5. Secondary Outcome: Clinical Attachment Level (CAL) Change Over Time (Mean CAL in All Subjects With Initial PD ≥ 4 mm) - Descriptive Statistics
Description: as for outcome 3
Time Frame: From baseline to 3 months and 6 months
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: millimeters
Groups:
- Other: Other Product Use Category - As Exposed Set
Arm/Group | IQOS | Cigarette | Dual User | Other
Number analyzed (Participants) | 70 | 84 | 17 | 1
millimeters
  Baseline: number analyzed (Participants) | 70 | 83 | 17 | 1
  Baseline | 4.65 [4.45 to 4.84] | 4.64 [4.45 to 4.82] | 4.60 [4.36 to 4.85] | 4.13
  Month 3 | 3.82 [3.57 to 4.07] | 3.79 [3.57 to 4.01] | 3.87 [3.48 to 4.26] | 3.20
  Month 6: number analyzed (Participants) | 69 | 83 | 17 | 1
  Month 6 | 3.74 [3.48 to 3.99] | 3.69 [3.46 to 3.91] | 3.64 [3.24 to 4.04] | 3.21

6. Secondary Outcome: Full-mouth Periodontal PD Change Over Time.
Description: Pocket depth (PD) is the distance from the gingival margin to which a probe penetrates into the pocket. Change in mean full-mouth PD will be measured, following mechanical periodontal therapy, in patients who switch to IQOS use compared to those who continue cigarette smoking.
Time Frame: From baseline to 3 months and 6 months
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: millimeters
Arm/Group | IQOS | Cigarette | Dual User | Other
Number analyzed (Participants) | 70 | 84 | 17 | 1
millimeters
  Baseline | 3.15 [3.02 to 3.29] | 3.20 [3.09 to 3.31] | 2.99 [2.80 to 3.17] | 2.92
  Month 3 | 2.70 [2.59 to 2.81] | 2.78 [2.67 to 2.88] | 2.69 [2.50 to 2.88] | 2.57
  Month 6: number analyzed (Participants) | 69 | 83 | 17 | 1
  Month 6 | 2.70 [2.58 to 2.82] | 2.72 [2.60 to 2.84] | 2.62 [2.39 to 2.84] | 2.55

7. Secondary Outcome: Full-mouth Clinical Attachment Level (CAL) Over Time.
Description: Clinical attachment level (CAL) is the measured distance from cementoenamel junction (CEJ) to the bottom of pocket using a periodontal probe. Change in mean full-mouth CAL will be measured, following mechanical periodontal therapy, in patients who switch to IQOS use compared to those who continue cigarette smoking.
Time Frame: From baseline to 3 months and 6 months
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: millimeters
Arm/Group | IQOS | Cigarette | Dual User | Other
Number analyzed (Participants) | 70 | 84 | 17 | 1
millimeters
  Baseline: number analyzed (Participants) | 70 | 83 | 17 | 1
  Baseline | 3.48 [3.26 to 3.69] | 3.52 [3.34 to 3.71] | 3.34 [3.00 to 3.69] | 2.99
  Month 3 | 3.10 [2.88 to 3.31] | 3.13 [2.93 to 3.32] | 3.15 [2.75 to 3.54] | 2.70
  Month 6: number analyzed (Participants) | 69 | 83 | 17 | 1
  Month 6 | 3.10 [2.86 to 3.33] | 3.09 [2.89 to 3.29] | 2.97 [2.59 to 3.36] | 2.70

8. Secondary Outcome: Peridontal PD Reduction.
Description: Pocket depth (PD) is the distance from the gingival margin to which a probe penetrates into the pocket. Mean PD change will be measured in sites with initial PD < 4 mm, and with initial PD of 4 mm to <5 mm, 5 mm to < 6 mm, 6 mm to < 7 mm and ≥ 7 mm.
Time Frame: From baseline to 3 months and 6 months
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: millimeters
Arm/Group | IQOS | Cigarette | Dual User | Other
Number analyzed (Participants) | 70 | 84 | 17 | 1
millimeters
  <4mm (Baseline) | 2.5 [2.5 to 2.6] | 2.6 [2.5 to 2.6] | 2.5 [2.4 to 2.6] | 2.6
  <4mm (Month 3: Change from Baseline) | -0.2 [-0.3 to -0.1] | -0.2 [-0.2 to -0.1] | -0.1 [-0.2 to 0.0] | -0.1
  <4mm (Month 6: Change from Baseline): number analyzed (Participants) | 69 | 83 | 17 | 1
  <4mm (Month 6: Change from Baseline) | -0.2 [-0.3 to -0.1] | -0.2 [-0.3 to -0.2] | -0.1 [-0.3 to 0.0] | -0.1
  4mm-5mm (Baseline) | 4.0 [4.0 to 4.0] | 4.0 [4.0 to 4.0] | 4.0 [4.0 to 4.0] | 4.0
  4mm-5mm (Month 3: Change from Baseline) | -0.8 [-0.9 to -0.7] | -0.8 [-0.9 to -0.7] | -0.8 [-0.9 to -0.6] | -1.0
  4mm-5mm (Month 6: Change from Baseline): number analyzed (Participants) | 69 | 83 | 17 | 1
  4mm-5mm (Month 6: Change from Baseline) | -0.9 [-1.0 to -0.8] | -0.9 [-1.0 to -0.8] | -0.8 [-1.1 to -0.6] | -0.9
  5mm-6mm (Baseline): number analyzed (Participants) | 65 | 80 | 17 | 1
  5mm-6mm (Baseline) | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0
  5mm-6mm (Month 3: Change from Baseline): number analyzed (Participants) | 65 | 80 | 17 | 1
  5mm-6mm (Month 3: Change from Baseline) | -1.2 [-1.3 to -1.0] | -1.1 [-1.2 to -0.9] | -1.0 [-1.3 to -0.7] | -1.8
  5mm-6mm (Month 6: Change from Baseline): number analyzed (Participants) | 70 | 79 | 17 | 1
  5mm-6mm (Month 6: Change from Baseline) | -1.2 [-1.4 to -1.0] | -1.2 [-1.4 to -1.1] | -1.2 [-1.6 to -0.9] | -2.0
  6mm-7mm (Baseline): number analyzed (Participants) | 48 | 59 | 14 | 1
  6mm-7mm (Baseline) | 6.0 [6.0 to 6.0] | 6.0 [6.0 to 6.0] | 6.0 [6.0 to 6.0] | NA — The sole subject in this use category did not have any sites with a PD ≥6mm.
  6mm-7mm (Month 3: Change from Baseline) | -1.3 [-1.6 to -1.0] | -1.2 [-1.4 to -0.9] | -1.4 [-2.0 to -0.8] | NA — The sole subject in this use category did not have any sites with a PD ≥6mm.
  6mm-7mm (Month 6: Change from Baseline): number analyzed (Participants) | 47 | 58 | 14 | 1
  6mm-7mm (Month 6: Change from Baseline) | -1.5 [-1.8 to -1.3] | -1.4 [-1.6 to -1.2] | -1.8 [-2.3 to -1.3] | NA — The sole subject in this use category did not have any sites with a PD ≥6mm.
  ≥7mm (Baseline): number analyzed (Participants) | 32 | 44 | 7 | 1
  ≥7mm (Baseline) | 7.6 [7.3 to 7.9] | 7.5 [7.3 to 7.6] | 8.4 [6.7 to 10.1] | NA — The sole subject in this use category did not have any sites with a PD ≥6mm.
  ≥7mm (Month 3: Change from Baseline): number analyzed (Participants) | 32 | 44 | 7 | 1
  ≥7mm (Month 3: Change from Baseline) | -2.1 [-2.5 to -1.6] | -1.6 [-2.0 to -1.1] | -2.5 [-3.6 to -1.3] | NA — The sole subject in this use category did not have any sites with a PD ≥6mm.
  ≥7mm (Month 6: Change from Baseline): number analyzed (Participants) | 32 | 43 | 7 | 1
  ≥7mm (Month 6: Change from Baseline) | -2.3 [-2.9 to -1.7] | -1.7 [-2.1 to -1.3] | -2.3 [-3.4 to -1.3] | NA — The sole subject in this use category did not have any sites with a PD ≥6mm.

9. Secondary Outcome: Clinical Attachment Level Improvement
Description: Clinical attachment level (CAL) is the measured distance from cementoenamel junction (CEJ) to the bottom of pocket using a periodontal probe. Mean CAL change will be measured in sites with initial PD < 4 mm, and with initial PD of 4 mm to <5 mm, 5 mm to < 6 mm, 6 mm to < 7 mm and ≥ 7 mm.
Time Frame: From baseline to 3 months and 6 months
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: millimeters
Arm/Group | IQOS | Cigarette | Dual User | Other
Number analyzed (Participants) | 70 | 84 | 17 | 1
millimeters
  <4mm (Baseline): number analyzed (Participants) | 70 | 83 | 17 | 1
  <4mm (Baseline) | 3.0 [2.8 to 3.1] | 3.0 [2.8 to 3.1] | 2.9 [2.6 to 3.3] | 2.6
  <4mm (Month 3: Change from Baseline) | -0.2 [-0.3 to -0.1] | -0.2 [-0.2 to -0.1] | 0.0 [-0.2 to 0.1] | -0.1
  <4mm (Month 6: Change from Baseline): number analyzed (Participants) | 69 | 82 | 17 | 1
  <4mm (Month 6: Change from Baseline) | -0.2 [-0.3 to 0.0] | -0.2 [-0.3 to -0.1] | -0.2 [-0.4 to 0.0] | -0.1
  4mm-5mm (Baseline): number analyzed (Participants) | 70 | 83 | 17 | 1
  4mm-5mm (Baseline) | 4.2 [4.1 to 4.4] | 4.2 [4.1 to 4.4] | 4.3 [4.1 to 4.6] | 4.1
  4mm-5mm (Month 3: Change from Baseline): number analyzed (Participants) | 70 | 83 | 17 | 1
  4mm-5mm (Month 3: Change from Baseline) | -0.7 [-0.8 to -0.6] | -0.7 [-0.8 to -0.6] | -0.6 [-0.8 to -0.4] | -0.9
  4mm-5mm (Month 6: Change from Baseline): number analyzed (Participants) | 69 | 82 | 17 | 1
  4mm-5mm (Month 6: Change from Baseline) | -0.8 [-0.9 to -0.6] | -0.8 [-0.9 to -0.7] | -0.8 [-1.0 to -0.5] | -0.9
  5mm-6mm (Baseline): number analyzed (Participants) | 65 | 79 | 17 | 1
  5mm-6mm (Baseline) | 5.2 [5.0 to 5.3] | 5.2 [5.0 to 5.3] | 5.2 [5.1 to 5.4] | 5.0
  5mm-6mm (Month 3: Change from Baseline): number analyzed (Participants) | 65 | 79 | 17 | 1
  5mm-6mm (Month 3: Change from Baseline) | -0.9 [-1.1 to -0.8] | -1.0 [-1.1 to -0.8] | -0.8 [-1.1 to -0.4] | -1.2
  5mm-6mm (Month 6: Change from Baseline): number analyzed (Participants) | 65 | 78 | 17 | 1
  5mm-6mm (Month 6: Change from Baseline) | -1.0 [-1.2 to -0.8] | -1.1 [-1.3 to -0.9] | -1.2 [-1.6 to -0.7] | -1.8
  6mm-7mm (Baseline): number analyzed (Participants) | 48 | 58 | 14 | 1
  6mm-7mm (Baseline) | 6.2 [6.0 to 6.5] | 6.3 [6.1 to 6.5] | 6.3 [6.0 to 6.6] | NA — The sole subject in this use category did not have any sites with a PD ≥6mm.
  6mm-7mm (Month 3: Change from Baseline): number analyzed (Participants) | 48 | 58 | 14 | 1
  6mm-7mm (Month 3: Change from Baseline) | -1.0 [-1.4 to -0.7] | -1.0 [-1.3 to -0.7] | -1.2 [-1.9 to -0.4] | NA — The sole subject in this use category did not have any sites with a PD ≥6mm.
  6mm-7mm (Month 6: Change from Baseline): number analyzed (Participants) | 47 | 57 | 14 | 1
  6mm-7mm (Month 6: Change from Baseline) | -1.3 [-1.6 to -0.9] | -1.3 [-1.5 to -1.0] | -1.7 [-2.2 to -1.2] | NA — The sole subject in this use category did not have any sites with a PD ≥6mm.
  ≥7mm (Baseline): number analyzed (Participants) | 32 | 43 | 7 | 1
  ≥7mm (Baseline) | 7.5 [6.9 to 8.1] | 7.9 [7.6 to 8.2] | 8.8 [6.4 to 11.2] | NA — The sole subject in this use category did not have any sites with a PD ≥6mm.
  ≥7mm (Month 3: Change from Baseline): number analyzed (Participants) | 32 | 43 | 7 | 1
  ≥7mm (Month 3: Change from Baseline) | -1.3 [-1.9 to -0.8] | -1.7 [-2.1 to -1.3] | -1.6 [-3.3 to 0.1] | NA — The sole subject in this use category did not have any sites with a PD ≥6mm.
  ≥7mm (Month 6: Change from Baseline): number analyzed (Participants) | 32 | 42 | 7 | 1
  ≥7mm (Month 6: Change from Baseline) | -1.6 [-2.2 to -0.9] | -1.9 [-2.2 to -1.5] | -2.0 [-4.0 to 0.1] | NA — The sole subject in this use category did not have any sites with a PD ≥6mm.

10. Secondary Outcome: Number of Periodontally Diseased Sites.
Description: Pocket depth (PD) is the distance from the gingival margin to which a probe penetrates into the pocket. Any change will be recorded in the number of periodontally diseased sites with Pocket Depth (PD) < 4 mm, with PD 4 mm to < 5mm, with PD 5 mm to < 6 mm , with PD 6 mm to < 7 mm and with PD ≥ 7 mm. PD is the distance from the gingival margin to which a probe penetrates into the pocket.
Time Frame: From baseline to 3 months and 6 months
Population: as for outcome 4
Measure: Number; unit: Number of sites
Arm/Group | IQOS | Cigarette | Dual User | Other
Number analyzed (Participants) | 70 | 84 | 17 | 1
Number of sites
  <4mm: Baseline | 7688 | 9194 | 1911 | 127
  <4mm: Month 3 | 9332 | 11146 | 2181 | 154
  <4mm: Month 6 | 9241 | 11199 | 2227 | 159
  4mm - 5mm: Baseline | 2067 | 2571 | 469 | 37
  4mm - 5mm: Month 3 | 1037 | 1393 | 261 | 14
  4mm - 5mm: Month 6 | 934 | 1241 | 259 | 8
  5mm - 6mm: Baseline | 724 | 1042 | 136 | 4
  5mm - 6mm: Month 3 | 366 | 483 | 102 | 0
  5mm - 6mm: Month 6 | 333 | 426 | 76 | 1
  6mm - 7mm: Baseline | 291 | 333 | 55 | 0
  6mm - 7mm: Month 3 | 151 | 238 | 31 | 0
  6mm - 7mm: Month 6 | 189 | 219 | 23 | 0
  ≥7mm: Baseline | 220 | 222 | 15 | 0
  ≥7mm: Month 3 | 124 | 113 | 10 | 0
  ≥7mm: Month 6 | 126 | 120 | 7 | 0
  Missing/Not done: Baseline | 26 | 12 | 0 | 0
  Missing/Not done: Month 3 | 6 | 1 | 1 | 0
  Missing/Not done: Month 6 | 7 | 1 | 0 | 0

11. Secondary Outcome: Gingival Inflammation
Description: Gingival inflammation will be measured by calculating the gingival index (GI) score for each target tooth.
  The gingival index (GI) scores each site on a 0 to 3 scale, with 0 being normal and 3 being severe inflammation characterized by edema, redness, swelling, and spontaneous bleeding.
Time Frame: From baseline to 3 months and 6 months
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: Gingival Index (GI)
Arm/Group | IQOS | Cigarette | Dual User | Other
Number analyzed (Participants) | 70 | 84 | 17 | 1
Gingival Index (GI)
  Baseline | 1.46 [1.35 to 1.57] | 1.48 [1.40 to 1.56] | 1.46 [1.28 to 1.64] | 1.38
  Month 3 | 1.06 [0.93 to 1.20] | 1.08 [0.97 to 1.19] | 1.22 [1.01 to 1.44] | 0.5
  Month 3: Change from Baseline | -0.40 [-0.52 to -0.28] | -0.40 [-0.51 to -0.29] | -0.24 [-0.44 to -0.03] | -0.88
  Month 6: number analyzed (Participants) | 69 | 83 | 17 | 1
  Month 6 | 1.03 [0.90 to 1.17] | 1.04 [0.93 to 1.15] | 1.05 [0.87 to 1.23] | 1.38
  Month 6: Change from Baseline: number analyzed (Participants) | 69 | 83 | 17 | 1
  Month 6: Change from Baseline | -0.43 [-0.55 to -0.30] | -0.44 [-0.56 to -0.31] | -0.41 [-0.67 to -0.15] | 0.00

12. Secondary Outcome: Tooth Mobility
Description: Tooth mobility will be graded according to Miller's mobility index (MMI), which is the most widely accepted method for routine clinical examinations of tooth mobility. The tooth is held between the metallic handles of two instruments and moved in the buccolingual or buccopalatal direction, and the moved distance is visually estimated by the person conducting the examination.
  Grade 0: Physiologic movement within 0.2 mm; Grade 1: Slight mobility, tooth can be moved 0.2 - 1 mm labiolingually; Grade 2: Moderate mobility, tooth can be moved 1 - 2 mm labiolingually or mesiodistally; Grade 3: Severe mobility, tooth can be moved more than 2 mm labiolingually or mesiodistally, or ability to depress the tooth in a vertical direction.
Time Frame: From baseline to 3 months and 6 months
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: MMI
Arm/Group | IQOS | Cigarette | Dual User | Other
Number analyzed (Participants) | 70 | 84 | 17 | 1
MMI
  Baseline | 0.18 [0.11 to 0.24] | 0.19 [0.12 to 0.26] | 0.23 [0.06 to 0.40] | 0
  Month 3 | 0.17 [0.10 to 0.24] | 0.16 [0.09 to 0.22] | 0.19 [0.03 to 0.34] | 0
  Month 3: Change from Baseline | -0.01 [-0.03 to 0.02] | -0.03 [-0.06 to -0.01] | -0.04 [-0.12 to 0.04] | 0.00
  Month 6: number analyzed (Participants) | 69 | 83 | 17 | 1
  Month 6 | 0.18 [0.10 to 0.26] | 0.17 [0.09 to 0.24] | 0.16 [0.04 to 0.27] | 0
  Month 6: Change from Baseline: number analyzed (Participants) | 69 | 83 | 17 | 1
  Month 6: Change from Baseline | 0.00 [-0.04 to 0.04] | -0.02 [-0.05 to 0.01] | -0.07 [-0.15 to 0.00] | 0.00

13. Secondary Outcome: Presence of Plaque on Tooth Surfaces in Full Mouth
Description: Plaque will be measured using the plaque control record (PCR) percentage.
Time Frame: From baseline to 3 months and 6 months
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: Plaque Control Record %
Arm/Group | IQOS | Cigarette | Dual User | Other
Number analyzed (Participants) | 70 | 84 | 17 | 1
Plaque Control Record %
  Baseline: number analyzed (Participants) | 69 | 84 | 17 | 1
  Baseline | 62.07 [57.68 to 66.46] | 62.48 [57.92 to 67.03] | 55.81 [44.62 to 67.99] | 77.68
  Month 3 | 48.03 [43.08 to 52.97] | 50.14 [45.66 to 54.62] | 44.56 [34.08 to 55.04] | 60.71
  Month 3: Change from Baseline: number analyzed (Participants) | 69 | 84 | 17 | 1
  Month 3: Change from Baseline | -14.27 [-19.04 to -9.49] | -12.34 [-15.70 to -8.99] | -11.25 [-21.45 to -1.05] | -16.96
  Month 6: number analyzed (Participants) | 69 | 83 | 17 | 1
  Month 6 | 49.60 [44.24 to 54.96] | 51.55 [47.20 to 55.90] | 47.92 [37.57 to 58.28] | 58.04
  Month 6: Change from Baseline: number analyzed (Participants) | 68 | 83 | 17 | 1
  Month 6: Change from Baseline | -13.27 [-18.14 to -8.41] | -11.22 [-14.72 to -7.71] | -7.89 [-17.75 to 1.98] | -19.64

14. Secondary Outcome: Inflammatory Status in Periodontal Pockets
Description: Gum inflammation was measured using percentage of teeth bleeding on probing (BOP).
  BOP in full mouth was measured to assess inflammatory status in the pocket and was assessed as YES or NO of bleeding at 6 sites per tooth. Gently probing (approximately 20 g pressure), the bleeding site within 30 seconds was assessed as YES.
Time Frame: From baseline to 3 months and 6 months
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: BOP %
Arm/Group | IQOS | Cigarette | Dual User | Other
Number analyzed (Participants) | 70 | 84 | 17 | 1
BOP %
  Baseline | 41.25 [35.94 to 46.56] | 42.93 [38.33 to 47.52] | 30.80 [23.96 to 37.65] | 48.81
  Month 3 | 26.68 [22.30 to 31.06] | 24.21 [20.70 to 27.71] | 19.03 [15.49 to 22.56] | 53.57
  Month 3: Change from Baseline | -14.57 [-19.03 to -10.11] | -18.72 [-21.84 to -15.60] | -11.78 [-16.48 to -7.07] | 4.76
  Month 6: number analyzed (Participants) | 69 | 83 | 17 | 1
  Month 6 | 26.90 [22.70 to 31.09] | 23.80 [20.10 to 27.50] | 19.80 [13.33 to 26.28] | 38.10
  Month 6: Change from Baseline: number analyzed (Participants) | 69 | 83 | 17 | 1
  Month 6: Change from Baseline | -14.85 [-19.16 to -10.54] | -18.71 [-22.33 to -15.10] | -11.00 [-16.83 to -5.17] | -10.71

15. Secondary Outcome: Concentrations of Urinary Nicotine Equivalents (NEQ)
Description: This biomarker of exposure to a tobacco smoke constituent will be measured in patients who switch to IQOS use and patients who continue cigarette smoking. Concentrations measured in urine and expressed as concentration adjusted for creatinine (mg/g creat).
Time Frame: From baseline to 3 months and 6 months
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: mg/g creat
Arm/Group | IQOS | Cigarette | Dual User | Other
Number analyzed (Participants) | 70 | 84 | 17 | 1
mg/g creat
  Baseline | 6.777 [5.625 to 8.165] | 7.649 [6.756 to 8.661] | 6.452 [3.935 to 10.580] | 8.527
  Month 3: number analyzed (Participants) | 70 | 83 | 17 | 1
  Month 3 | 6.766 [5.611 to 8.158] | 6.699 [5.620 to 7.986] | 5.911 [3.820 to 9.146] | 7.681
  Month 6: number analyzed (Participants) | 68 | 83 | 17 | 1
  Month 6 | 6.471 [5.235 to 7.999] | 6.563 [5.337 to 8.071] | 5.467 [3.044 to 9.816] | 5.213

16. Secondary Outcome: Concentrations of Total 4-(Methylnitrosamino)-1-(3-pyridyl)-1-butanol (Total NNAL)
Description: This biomarker of exposure to a tobacco smoke constituent will be measured in patients who switch to IQOS use and patients who continue cigarette smoking. Concentrations measured in urine and expressed as concentration adjusted for creatinine (pg/mg creat).
Time Frame: From baseline to 3 months and 6 months
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: pg/mg creat
Arm/Group | IQOS | Cigarette | Dual User | Other
Number analyzed (Participants) | 70 | 84 | 17 | 1
pg/mg creat
  Baseline | 83.30 [65.33 to 106.20] | 112.52 [92.19 to 137.35] | 93.01 [58.11 to 148.84] | 159.05
  Mionth 3: number analyzed (Participants) | 70 | 83 | 17 | 1
  Mionth 3 | 25.77 [20.03 to 33.16] | 100.67 [80.95 to 125.20] | 68.62 [39.17 to 120.23] | 124.39
  Month 6: number analyzed (Participants) | 68 | 83 | 17 | 1
  Month 6 | 22.55 [17.28 to 29.45] | 96.70 [75.97 to 123.09] | 77.17 [45.80 to 130.03] | 48.74

17. Secondary Outcome: Concentrations of 2-cyanoethylmercapturic Acid (CEMA)
Description: This biomarker of exposure to a tobacco smoke constituent will be measured in patients who switch to IQOS use and patients who continue cigarette smoking. Concentrations measured in urine and expressed as concentration adjusted for creatinine (ng/mg creat).
Time Frame: From baseline to 3 months and 6 months
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mg creat
Arm/Group | IQOS | Cigarette | Dual User | Other
Number analyzed (Participants) | 70 | 84 | 17 | 1
ng/mg creat
  Baseline | 67.29 [52.25 to 86.67] | 90.44 [74.00 to 110.54] | 92.10 [59.04 to 143.66] | 140.95
  Month 3: number analyzed (Participants) | 70 | 83 | 17 | 1
  Month 3 | 9.94 [7.35 to 13.43] | 80.30 [63.38 to 101.74] | 50.36 [27.16 to 93.41] | 5.19
  Month 6: number analyzed (Participants) | 68 | 83 | 17 | 1
  Month 6 | 7.56 [5.53 to 10.33] | 76.65 [59.37 to 98.97] | 69.02 [37.51 to 127.01] | 1.97

18. Secondary Outcome: Use of Tobacco or Nicotine-containing Products in Patients Switching to IQOS Use and Patients Who Continue Cigarette Smoking.
Description: Self-reported use of tobacco or nicotine containing products will be measured over the study in patients switching to IQOS use and patients who continue cigarette smoking.
Time Frame: From baseline to 6 months
Population: The analysis population consisted of all randomized subjects with at least one product use experience and at least one valid non-safety assessment analyzed by actual product use. Results were reported only for subjects with exposure to a specific tobacco or nicotine-containing product.
Measure: Mean (95% Confidence Interval); unit: number of product units consumed
Arm/Group | IQOS | Cigarette | Dual User | Other
Number analyzed (Participants) | 70 | 84 | 17 | 1
number of product units consumed
  Cigarettes/day over the last five years (Baseline) | 18.2 [16.7 to 19.7] | 17.7 [16.6 to 18.9] | 18.1 [15.1 to 21.1] | 20.0
  Cigarettes/day: number analyzed (Participants) | 21 | 84 | 17 | 0
  Cigarettes/day | 0.22 [0.10 to 0.34] | 17.06 [15.77 to 18.35] | 8.16 [3.58 to 12.73] |
  IQOS Heatsticks/day: number analyzed (Participants) | 70 | 2 | 17 | 0
  IQOS Heatsticks/day | 16.60 [15.19 to 18.02] | 0.30 [0.00 to 3.51] | 9.06 [6.86 to 11.25] |
  Other Heat-Not-Burn/day: number analyzed (Participants) | 1 | 3 | 2 | 1
  Other Heat-Not-Burn/day | 1.67 | 3.72 [0.00 to 14.24] | 0.01 [0.00 to 0.04] | 30.00
  E-cigarettes/day: number analyzed (Participants) | 1 | 0 | 0 | 0
  E-cigarettes/day | 2.67 |  |  |
  Nicotine Replacement Therapy/day: number analyzed (Participants) | 0 | 1 | 0 | 1
  Nicotine Replacement Therapy/day |  | 0.81 |  | 0.50

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the signature of the ICF by each subject until the end of the safety follow-up period, for a total study duration of up to 31 weeks for each subject.
Description: The safety population comprised the 179 subjects enrolled in the study, of which 172 subjects were randomized to the IQOS or Cigarette arms.
  Adverse events are reported according to subjects' product exposure over the study period (Product Use Category, i.e., IQOS use; Cigarette use; Dual use; or Other use) as detailed in the "Arm/Group" (Reporting Groups) table.
  The seven subjects who were enrolled but not randomized are included in the Cigarette group for adverse event reporting.
Groups:
- IQOS: IQOS users (safety population)
- Cigarette: Cigarette users (safety population; includes 7 subjects who were enrolled but not randomized and were considered to be in the cigarette users group)
- Dual: Dual users (safety population)
- Other: Other users (safety population)
Arm/Group | IQOS | Cigarette | Dual | Other
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/91 | 0/17 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/70 | 2/91 | 0/17 | 0/1
Other Adverse Events (participants affected / at risk) | 25/70 | 29/91 | 13/17 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IQOS (N=70) | Cigarette (N=91) | Dual (N=17) | Other (N=1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Jaw cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IQOS (N=70) | Cigarette (N=91) | Dual (N=17) | Other (N=1)
Dental caries (Gastrointestinal disorders) | 6 (6) | 12 (12) | 3 (3) | 0 (0)
Toothache (Gastrointestinal disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 8 (8) | 5 (5) | 2 (2) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Procedural Pain (Injury, poisoning and procedural complications) | 1 (1) | 4 (4) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperaesthesia (Nervous system disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Device breakage (Product Issues) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device failure (Product Issues) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Gingival Pain (Gastrointestinal disorders) | 2 (2) | 3 (3) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gingivitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
We confirm we have the contractual provisions in place which specify that in no event will the study site be allowed to disclose to any third party (or publicly release) any information obtained through the study without the CRO's prior written consent which in turn cannot provide such consent without Sponsor's approval unless such publication is made to satisfy regulatory requirements.

The Intellectual Property rights and research results from the present study belong to the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2019-01-09): https://cdn.clinicaltrials.gov/large-docs/51/NCT03364751/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-07): https://cdn.clinicaltrials.gov/large-docs/51/NCT03364751/SAP_001.pdf